CLINICAL TRIAL: NCT00679198
Title: Improving Osteoporosis Care in High-Risk Home Health Patients Through a High-Intensity Intervention
Brief Title: Improving Osteoporosis Care in High-Risk Home Health Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Alacare Home Health and Hospice (Other)
Responsible Party: Principal Investigator, Meredith Kilgore, PhD, RN, Associate Professor of Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: X071029007
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Patient Compliance; Communication; Osteoporosis; Fractures, Bone
Keywords: osteoporosis; fracture; communication; prescription medication
MeSH Terms: conditions — Patient Compliance; Communication; Osteoporosis; Fractures, Bone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): We will train home health nurses to act as patient advocates by communicating the risks and benefits of osteoporosis treatment to patients and their healthcare providers
  Interventions: Behavioral: nurse-patient communication
- 2 (No Intervention): Standard care

INTERVENTIONS:
Behavioral: nurse-patient communication — We will train home health nurses to act as patient advocates by communicating the risks and benefits of osteoporosis treatment to patients and their healthcare providers.
  Thus, we will provide a comprehensive, integrated approach to the management of osteoporosis among patients with a history of insufficiency fractures that is highly generalizable to a national setting.
  Arms: 1

SUMMARY:
SPECIFIC AIMS: We propose a three-year study to develop a high-intensity intervention to improve osteoporosis care and test a novel intervention in a group-randomized trial of 27 home health offices and 1,000 patients referred to home health care with a history of fracture.

Aim 1. Develop an intervention to promote osteoporosis treatment that includes: (1) training to enhance nurse-patient and nurse-physician risk communication regarding osteoporosis and fracture risk; (2) automated prompts within the home health agency's electronic medical record system to promote appropriate osteoporosis management; and (3) implementation of osteoporosis-related standardized care pathways and order sets.

Aim 2. Conduct a group-randomized trial to test the effectiveness of the intervention to promote initial use of osteoporosis medications and adherence to treatment after discharge from home health. We hypothesize that:

H1: Patients in the intervention group will have increased initial receipt of osteoporosis prescription medications and calcium/vitamin D supplements to prevent and treat osteoporosis compared to patients receiving usual care; H2: Patients in the intervention group will demonstrate increased persistence in the use of these therapies compared to those receiving usual care.

Secondary Aims (SA) will include exploratory analyses of fracture related morbidity and mortality, patient-reported quality of life, and health services utilization and costs.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be identified as "at-risk" if they are referred to home health care for post-fracture care or if they are admitted for another reason and have a previous diagnosis of fracture.

Exclusion Criteria:

* Patients in hospice, with a life expectancy < 1 year, over 95 years old, or with concomitant metabolic bone diseases (e.g. Paget's disease of bone) will be excluded.

Max Age: 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 667 (Actual)
Dates: Start 2009-03; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Increased receipt of osteoporosis prescription medications and calcium/vitamin D supplements to prevent and treat osteoporosis | within 3 months of discharge from home health care

SECONDARY OUTCOMES:
Increased persistence in the use of these therapies | 18 months after their discharge from home health care

CONTACTS AND LOCATIONS:
Overall Officials: Meredith L Kilgore, PhD RN, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham Department of Rheumatology, Birmingham, Alabama, United States